CLINICAL TRIAL: NCT00435552
Title: Ease-it Spray for the Treatment of Fire Ant Stings
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: C.R.Darnall Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: C.2007.001
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2007-02-15 (Estimated); Status verified 2007-01

CONDITIONS: Insect Bites and Stings
MeSH Terms: conditions — Insect Bites and Stings

INTERVENTIONS:
Procedure: Ease-It Spray

SUMMARY:
The application of Ease-it Spray will alleviate pain secondary to fire ant stings more quickly than placebo.

ELIGIBILITY:
Inclusion Criteria:

* AD soldier in US Army
* Ages 18-60
* Volunteer
* Absence of serious medical condition
* Past allergic reactions
* Asthma
* History of (h/o) IFA sting

Exclusion Criteria:

* Inability to provide informed consent
* Known h/o hymenoptera allergic reaction
* Allergy to any component of the treatments
* Inability to follow-up
* Active medical condition
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Dates: Start 2007-02